CLINICAL TRIAL: NCT05620953
Title: Severe Acute Respiratory Infections Surveillance in Belgium (2011-2020, Prior to COVID-19 Pandemic)
Brief Title: Severe Acute Respiratory Infections (SARI) in Belgium (2011-2020)
Acronym: SARIpreSC2
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Collaborators: Belgian Federal Public Service, Food Chain Safety and Environment (Other Government); Centre Hospitalier Universitaire Saint Pierre (Other); AZ Sint-Jan AV (Other); Universitair Ziekenhuis Brussel (Other); Grand Hôpital de Charleroi (Other); Jessa Hospital (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Principal Investigator, Cyril Barbezange, scientist, Sciensano
Other Study IDs: SARI-11-20
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Influenza Viral Infections; Respiratory Viral Infection; Severe Acute Respiratory Infection
Keywords: sentinel surveillance
MeSH Terms: interventions — Respiratory Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — respiratory specimens (mainly nasopharyngeal swabs, but a few nasal aspirates and broncho-alveolar lavages)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARI case
  Interventions: Diagnostic Test: respiratory specimen

INTERVENTIONS:
Diagnostic Test: respiratory specimen — nasopharyngeal swab or nasal aspiration or broncho-alveolar lavage

SUMMARY:
The Belgian Severe Acute Respiratory Infections network (BELSARI-net) was implemented during the influenza season 2011-2012 following the recommendations of the World Health Organization (WHO) to monitor severity of influenza viruses in hospitals. The network is composed of 6 hospitals throughout the country, two in each administrative region (Flanders, Wallonia and Brussels-Capital), and operates during the influenza epidemic period (from the last week of December or first/second week of January to the third/last week of April, depending on when influenza virus circulation is detected by the general population, based on the Influenza-like illness (ILI) network of general practitioners).

Enrollment is performed for all cases matching the SARI case definition (based on WHO's case definition) and accepting to take part. A respiratory specimen is sampled systematically from each participant, and detailed clinico-epidemiological data, such as information on age, sex, symptoms and potential risk factors such as pregnancy or comorbidities (chronic respiratory diseases, asthma, chronic cardiovascular diseases, renal insufficiency, obesity, diabetes, hepatic or renal insufficiency, immunodeficiency, neuromuscular disease, pregnancy) is also collected. Participants are followed up during hospitalization for the occurrence of complications (detection of pneumonia based on chest radiography, development of acute respiratory distress syndrome (ARDS), requirement for respiratory assistance and/or for extracorporeal membrane oxygenation (ECMO), admission in intensive care unit (ICU)), or death (all-cause death).

The current project includes all the samples received by the Belgian National Influenza Centre (NIC) during the influenza seasons 2011-2012 till 2019-2020.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric and adult patients admitted to one of the 6 sentinel hospitals during the active surveillance and fulfilling the case definition of acute respiratory infection with onset within the last ten days, with history of fever or measured fever of ≥38°C, with cough and/or dyspnea, and overnight hospitalization.

Exclusion Criteria:

* nosocomial infection, i.e. symptoms appearing after admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to one of the 6 participating hospital during the season surveillance dates.
Sampling Method: Non-Probability Sample
Enrollment: 12145 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Number of participants positive for influenza viruses | within 10 days after symptom onset
  result of influenza PCR detection test (typing and subtyping)
Number of participants positive for non-influenza viruses | within 10 days after symptom onset (only routinely tested since influenza season 2015-2016)
  results of non-influenza multiplex PCR detection test (16 targets)
Number of participants who died during hospitalization | from date of hospital admission until date of death during hospitalization or date of hospital exit
  alive or dead

SECONDARY OUTCOMES:
Number of participants with at least one known risk factor | on date of hospital admission
  existence of co-morbidities or known risk factors among a list provided on form
Number of participants who experienced at least one complication | from date of hospital admission until date of death during hospitalization or date of hospital exit
  occurence of complications (among a list provided on form) during hospitalisation stay

REFERENCES:
- [Result] Subissi L, Bossuyt N, Reynders M, Gerard M, Dauby N, Lacor P, Daelemans S, Lissoir B, Holemans X, Magerman K, Jouck D, Bourgeois M, Delaere B, Quoilin S, Van Gucht S, Thomas I, Barbezange C. Spotlight influenza: Extending influenza surveillance to detect non-influenza respiratory viruses of public health relevance: analysis of surveillance data, Belgium, 2015 to 2019. Euro Surveill. 2021 Sep;26(38):2001104. doi: 10.2807/1560-7917.ES.2021.26.38.2001104. PMID 34558405
- [Result] Fischer N, Dauby N, Bossuyt N, Reynders M, Gerard M, Lacor P, Daelemans S, Lissoir B, Holemans X, Magerman K, Jouck D, Bourgeois M, Delaere B, Quoilin S, Van Gucht S, Thomas I, Barbezange C, Subissi L. Monitoring of human coronaviruses in Belgian primary care and hospitals, 2015-20: a surveillance study. Lancet Microbe. 2021 Mar;2(3):e105-e114. doi: 10.1016/S2666-5247(20)30221-4. Epub 2021 Jan 27. PMID 33937883
- [Result] Subissi L, Bossuyt N, Reynders M, Gerard M, Dauby N, Bourgeois M, Delaere B, Quoilin S, Van Gucht S, Thomas I, Barbezange C. Capturing respiratory syncytial virus season in Belgium using the influenza severe acute respiratory infection surveillance network, season 2018/19. Euro Surveill. 2020 Oct;25(39):1900627. doi: 10.2807/1560-7917.ES.2020.25.39.1900627. PMID 33006303
- [Result] Fischer N, Moreels S, Dauby N, Reynders M, Petit E, Gerard M, Lacor P, Daelemans S, Lissoir B, Holemans X, Magerman K, Jouck D, Bourgeois M, Delaere B, Quoilin S, Van Gucht S, Thomas I, Bossuyt N, Barbezange C. Influenza versus other respiratory viruses - assessing severity among hospitalised children, Belgium, 2011 to 2020. Euro Surveill. 2023 Jul;28(29):2300056. doi: 10.2807/1560-7917.ES.2023.28.29.2300056. PMID 37470740